CLINICAL TRIAL: NCT01799811
Title: Prospective, Multicenter, Primary Below the Knee Bypass Evaluation With CryoVein® Cryopreserved Saphenous Vein Allograft in Patients With Critical Limb Ischemia
Brief Title: Cryopreserved Saphenous Vein Allograft in Patients With Critical Limb Ischemia for Peripheral Revascularization
Acronym: LIMBSAVE
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: Artivion Inc. (Industry)
Other Study IDs: AVG1201.000-M
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
Keywords: allograft; limb salvage; patency; Cryopreserved; open bypass
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the Study follow-up period, a patient may present with an event requiring an open surgical revision, surgical explant or limb amputation on the (allograft) recipient limb. At the time of related planned intervention a tissue sample of the affected area of the allograft may be obtained and, if so, will placed into 10% buffered formalin solution and returned to CryoLife for histologic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CLI patient's needing open bypass: Patients presenting with Rutherford Class 5 or 6 CLI that are being evaluated for open peripheral arterial revascularization.

SUMMARY:
The objective Study is to evaluate the short- and long-term clinical outcomes of patients receiving the CryoVein cryopreserved saphenous vein allograft (CVA) as their primary open bypass conduit to assess if there is a quantifiable correlation to time of placement as a primary bypass graft and improved long-term clinical outcomes of patients with critical limb ischemia (CLI).

DETAILED DESCRIPTION:
A minimum of 50 CVA will be implanted in enrolled patients at up to 6 participating sites. The Study will include prospective evaluations on these patients at discharge, 1, 3, 6, 9, 12, 18 and 24 months following surgery. The window for follow-up visits is ± 2 weeks for each time point. All Study patients will be expected to participate in all follow-up evaluations unless precluded by patient death.

Patient status and graft performance data will be collected on all patients consented and enrolled into the Study. The primary endpoint of the Study will be limb salvage. The secondary endpoints of the Study will include primary patency, secondary patency, morbidity and mortality per the same reporting standards.

Patient attributes (age, gender, etc.) and preoperative assessments (indication for surgery, medical history) will be summarized using descriptive statistics. Graft performance will be presented as freedom from an event endpoint (patient death, graft complication, amputation, graft explant) as calculated by the Kaplan-Meier method. Log Rank and Cox Regression will be utilized for comparison between subgroups of the patient population. Statistical software will be used to compile and analyze all submitted clinical data.

The method of data reporting may include, but is not limited to, a description of the sample population, frequency distributions of patient demographics, allograft statistics, and follow-up percentages, summary of event data, correlation analysis, and actuarial analysis

ELIGIBILITY:
Inclusion Criteria:

* Patient is an acceptable candidate to receive primary open bypass on the limb receiving the CVA.
* CLI diagnosis of Rutherford Class 5 or 6.
* Tibio-peroneal trunk, Tibial or Peroneal outflow artery.
* Minimum of 1 patent run-off artery.
* Serum Creatinine < 2.4 mg/dl.
* Life expectancy > 2 years from consent.
* 18 years of age or older at the time of consent.
* Male or non-pregnant female.
* Ability to understand and provide written informed consent.
* Willing and able to attend and cooperate with the follow-up examinations.
* Able to follow Study required post-operative daily aspirin and/or other oral anticoagulation/antiplatelet regimen.

Exclusion Criteria:

* Patient currently receiving hemodialysis for end stage renal disease.
* Known hypercoaguable state.
* Known heparin allergy.
* Patients with any condition which, in the opinion of the investigator could preclude evaluation of response or completion of follow-up or affect patient safety.
* Currently being treated with an investigational device or drug (within 3 months prior to surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with Rutherford Class 5 or 6 CLI that are being evaluated for open peripheral arterial revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Limb Salvage | Assessed for 24 months following surgery.
  Patients will undergo follow-up assessment for limb salvage.

SECONDARY OUTCOMES:
Patency | Assessed until graft failure over a period of 24 months. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months".
  Patients with functional grafts will undergo follow-up Study evaluation via Duplex Ultrasound.

OTHER OUTCOMES:
All cause morbidity and mortality | Assessed for 24 months following implant surgery.
  Data will be collected on any graft complications such as, but not limited to occlusion, bleeding complications, infection, or aneurysm. Patient survival will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (7):
- United States (7):
  - Arizona Heart Institue, Phoenix, Arizona
  - Veteran's Administration, Palo Alto, California
  - University of California at San Francisco, San Francisco, California
  - Sacred Heart Hospital, Pensacola, Florida
  - Carle Foundation Hospital, Urbana, Illinois
  - University of Texas Medical Branch, Galveston, Texas
  - Scott & White Memorial Hospital, Temple, Texas

IPD SHARING:
Plan to Share IPD: No
Post market study of 361 product; not supporting any FDA approvals.

REFERENCES:
- [Background] Walker PJ, Mitchell RS, McFadden PM, James DR, Mehigan JT. Early experience with cryopreserved saphenous vein allografts as a conduit for complex limb-salvage procedures. J Vasc Surg. 1993 Oct;18(4):561-8; discussion 568-9. PMID 8411463
- [Background] Shah RM, Faggioli GL, Mangione S, Harris LM, Kane J, Taheri SA, Ricotta JJ. Early results with cryopreserved saphenous vein allografts for infrainguinal bypass. J Vasc Surg. 1993 Dec;18(6):965-9; discussion 969-71. doi: 10.1067/mva.1993.50617. PMID 8264053
- [Background] Leseche G, Penna C, Bouttier S, Joubert S, Andreassian B. Femorodistal bypass using cryopreserved venous allografts for limb salvage. Ann Vasc Surg. 1997 May;11(3):230-6. doi: 10.1007/s100169900039. PMID 9140596
- [Background] Martin RS 3rd, Edwards WH, Mulherin JL Jr, Edwards WH Jr, Jenkins JM, Hoff SJ. Cryopreserved saphenous vein allografts for below-knee lower extremity revascularization. Ann Surg. 1994 Jun;219(6):664-70; discussion 670-2. doi: 10.1097/00000658-199406000-00009. PMID 8203975
- [Background] Farber A, Major K, Wagner WH, Cohen JL, Cossman DV, Lauterbach SR, Levin PM. Cryopreserved saphenous vein allografts in infrainguinal revascularization: analysis of 240 grafts. J Vasc Surg. 2003 Jul;38(1):15-21. doi: 10.1016/s0741-5214(03)00330-6. PMID 12844083
- [Background] Bannazadeh M, Sarac TP, Bena J, Srivastava S, Ouriel K, Clair D. Reoperative lower extremity revascularization with cadaver vein for limb salvage. Ann Vasc Surg. 2009 Jan-Feb;23(1):24-31. doi: 10.1016/j.avsg.2008.04.011. Epub 2008 Jul 26. PMID 18657383
- [Background] Buckley CJ, Abernathy S, Lee SD, Arko FR, Patterson DE, Manning LG. Suggested treatment protocol for improving patency of femoral-infrapopliteal cryopreserved saphenous vein allografts. J Vasc Surg. 2000 Oct;32(4):731-8. doi: 10.1067/mva.2000.110049. PMID 11013037
- [Background] Zehr BP, Niblick CJ, Downey H, Ladowski JS. Limb salvage with CryoVein cadaver saphenous vein allografts used for peripheral arterial bypass: role of blood compatibility. Ann Vasc Surg. 2011 Feb;25(2):177-81. doi: 10.1016/j.avsg.2010.07.020. PMID 20889296
- [Background] Randon C, Jacobs B, De Ryck F, Beele H, Vermassen F. Fifteen years of infrapopliteal arterial reconstructions with cryopreserved venous allografts for limb salvage. J Vasc Surg. 2010 Apr;51(4):869-77. doi: 10.1016/j.jvs.2009.11.062. PMID 20347683